CLINICAL TRIAL: NCT04246320
Title: Taking Brain Monitoring to the Next Level
Acronym: HDBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Rajesh Kumar, PhD, Professor In-Residence, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HDBRAIN 16-001040
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium; Obstructive Sleep Apnea
Keywords: goal directed therapy (GDT); magnetic resonance imaging (MRI); neurocognitive testing
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium; Sleep Apnea, Obstructive | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): Patients monitored and receiving a standard anesthesia plan in addition of a goal directed therapy (GDT) hemodynamic management (MAP > 60 mmHg) and processed EEG-guided anesthesia (PSI targeted between 30-50).
  Interventions: Other: Goal directed therapy (GDT)

INTERVENTIONS:
Other: Goal directed therapy (GDT) — Goal directed therapy (GDT) hemodynamic management (MAP > 60 mmHg) and processed EEG-guided anesthesia (PSI targeted between 30-50).

SUMMARY:
This one arm clinical study will assess the impact of a goal directed therapy intervention, aiming at optimizing depth of anesthesia and intraoperative blood pressure on the incidence of postoperative cognitive dysfunction and delirium relative to a standardized anesthetic plan. We will enroll 60 patients and will measure the neurocognitive status (MoCA test) of patients before and after surgery (at discharge, within 2 weeks after surgery and 6 months after surgery) to determine the relative impact of anesthetic care on the development of postoperative delirium and cognitive decline. All patients will have a brain scan (fMRI) before and after surgical intervention. Patients will also be asked to participate in an optional blood draw which will take place during their brain imaging visit and post operatively (within 2 days after surgery).

DETAILED DESCRIPTION:
This study will test the hypothesis that a goal directed therapy intervention, which optimizes depth of anesthesia and intraoperative blood pressure can decrease the incidence of postoperative neurocognitive dysfunction

Subjects will be recruited for the study and the protocol explained. In addition to standard American Society of Anesthesiologists (ASA) monitoring, we will monitor continuous non-invasive blood pressure and 4 lead electroencephalogram (EEG) channels. Patients will receive standardized anesthesia care in addition to a goal directed therapy hemodynamic management (MAP > 60 mmHg) and processed EEG-guided anesthesia (PSI targeted between 30-50).

Neurocognitive testing: In order to assess general cognitive function, the Montreal Cognitive Assessment test will be used. Cognitive function will be measured preoperatively and postoperatively at discharge, 1 month and 6 months after surgery. For delirium measurement, we will administer daily the Confusion Assessment Method (CAM-ICU) for up to 3 days.

The Montreal Cognitive Assessment (MoCA) is a screening tool to assess mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructionals skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.

The Wide Range Assessment of Memory and Learning (WRAML2) is a broad-based memory battery that provides a flexible measure of memory functioning and learning and takes approximately 45-60 minutes to administer. This assessment will be conducted at the first MRI visit and at the 6 month follow up.

The Confusion Assessment Method for the ICU (CAM-ICU) screens for the development of delirium and assesses four features: 1) acute change or fluctuation in mental status from baseline, 2) inattention, 3) altered level of consciousness, and 4) disorganized thinking. The CAM-ICU is positive, and the patient is considered to have delirium, if features 1 and 2 and either feature 3 or 4 are present.

Brain imaging: The timing of pre-operative brain imaging will be as allowed by patient factors and scanner availability, typically less than 15 days before surgery, when the patient comes for the preoperative evaluation, and postoperatively within 2 weeks after surgery.

Optional Blood Draws: Patients will be asked to provide 2 optional blood samples, drawn the day of their brain imaging visit and post-operatively (within 2 days). These samples will be used to asses blood inflammatory biomarkers in obstructive sleep apnea (OSA) subjects and non-OSA subjects between baseline and post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* 45-75 years old,
* undergoing abdominal, orthopedic, gynecological, or urological surgery
* expected to stay in hospital for at least 24hours

Exclusion Criteria:

* Substantial hearing impairment or inability to understand English, since there needs to be neurocognitive testing done
* status post craniotomy
* severe dementia

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-08-13 (Actual)

PRIMARY OUTCOMES:
Postoperative cognitive dysfunction | Preoperatively (within 15 days of surgery)
  Montreal Cognitive Assessment (MoCA) test
Postoperative cognitive dysfunction | postoperatively at discharge (within 2 weeks of surgery).
  Montreal Cognitive Assessment (MoCA) test
Postoperative cognitive dysfunction | 6 months after surgery.
  Montreal Cognitive Assessment (MoCA) test
Postoperative Delirium | Daily for up to 3 days postoperatively
  Confusion Assessment Method (CAM-ICU)

SECONDARY OUTCOMES:
Examining brain changes | Typically less than 15 days before surgery, when the patient comes for the preoperative evaluation, postoperatively at up to 48 hours after surgery, and 6 months post surgery
  Using non-invasive magnetic resonance imaging based diffusion tensor imaging
Examining brain changes II | postoperatively within 2 weeks of surgery
  Using non-invasive magnetic resonance imaging based diffusion tensor imaging
Examining brain changes III | 6 months post surgery
  Using non-invasive magnetic resonance imaging based diffusion tensor imaging
Blood anti-inflammatory biomarkers | pre-operatively (within 15 days before surgery)
  Assess blood inflammatory biomarkers (Il6, Il10, TNFa, IL1b, HMGB1) in OSA subjects and non-OSA subjects
Blood anti-inflammatory biomarkers | post-operatively (within 2 days of surgery)
  Assess blood inflammatory biomarkers (Il6, Il10, TNFa, IL1b, HMGB1) in OSA subjects and non-OSA subjects

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Kumar, PhD, Principal Investigator — University of California, Los Angeles; Susana Vacas, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology & Perioperative Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joosten A, Rinehart J, Bardaji A, Van der Linden P, Jame V, Van Obbergh L, Alexander B, Cannesson M, Vacas S, Liu N, Slama H, Barvais L. Anesthetic Management Using Multiple Closed-loop Systems and Delayed Neurocognitive Recovery: A Randomized Controlled Trial. Anesthesiology. 2020 Feb;132(2):253-266. doi: 10.1097/ALN.0000000000003014. PMID 31939839
- [Background] Vacas S, Cannesson M. Noninvasive Monitoring and Potential for Patient Outcome. J Cardiothorac Vasc Anesth. 2019 Aug;33 Suppl 1(Suppl 1):S76-S83. doi: 10.1053/j.jvca.2019.03.045. No abstract available. PMID 31279357